CLINICAL TRIAL: NCT03501563
Title: Effects of Hypotensive Anesthesia on Thiol Disulphide Balance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Leyla Kazancıoğlu, Assistant Professor, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 2018/63
Record Dates: First submitted 2018-04-06; First posted 2018-04-18 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Nasal Septum Deviation
Keywords: hypotensive anesthesia; thiol / disulfide; oxidative stress markers; septoplasty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Case Group: Participants with ASA 1-2, aged 18-60 years, undergoing hypotensive anesthesia in the operation of the septoplasty in Recep Tayyip Erdoğan University Medical Faculty Training and Research Hospital. Participants with uncontrolled hypertension, diabetes mellitus, cerebrovascular disease, cogulopathy, morbid obesity (BMI ≥35) and renal disease will not be taken.
  Participants were first pre-medicated with an infusion of midazolam 0.05 mg/kg, fentanyl 1 µg/kg, lidocaine 1 mg/kg. Induction of anesthesia was achieved with an infusion of propofol 1-2 mg/kg and vecuronium bromide 0.6 mg/kg and after 2 to 3 minutes participants were intubated with the appropriate tube size. Anesthesia was maintained with an infusion of remi fentanyl (0.05 - 1 µg/Kg/min), with oxygen (O2) in air with desflurane.

SUMMARY:
Oxidative stress at the cellular level and the effects of the antioxidant system on the anesthetic drugs make the anesthesia method more important. Hypotensive anesthesia or controlled hypotension is an anesthetic technique routinely used in many operations (ENT, orthopedic, plastic surgery, etc.) to reduce intraoperative bleeding and to provide a more open surgical area.

In this study, investigators aimed to investigate the effects of hypotensive anesthesia on thiol / disulfide balance from oxidative stress markers.

Hypotensive anesthesia is caused by hypoperfusion and hypoxia-induced oxidative stresses at the tissue level and can initiate cell damage. Many methods can be used alone or in combination to create hypotensive anesthesia. İnvestigators will investigate whether hypotensive anesthesia causes an effect on the cellular level.

DETAILED DESCRIPTION:
This study will be performed prospectively with 80 participants with ASA 1-2, aged 18-60 years, undergoing hypotensive anesthesia in the operation of the septoplasty in Recep Tayyip Erdoğan University Medical Faculty Training and Research Hospital. Participants with uncontrolled hypertension, diabetes mellitus, cerebrovascular disease, cogulopathy, morbid obesity (BMI ≥35) and renal disease will not be taken. Anesthesia induction and management will be standardized. Hypotension in the participants will be maintained by reducing the mean arterial pressure (MAP) by 30% or 55-65 mmHg according to the initial value. In the study, the heart rate (HR), MAP, peripheral O2 saturation (SpO2), ETCO2 (end-tidal carbon dioxide) values, and BIS (Bispectral index) values showing anesthesia depth are to be followed. Participants will receive venous blood sample of up to 2 ml before the anesthesia induction and 10 minutes to finish of the hypotensive anesthesia, from the untreated vein. Thiol disulfide levels from this blood sample will be studied in the biochemistry research laboratory using the method developed by Erel et al.

ELIGIBILITY:
Inclusion Criteria:

(American Society of Anesthesiologists) ASA Classification I - II controlled hypotensive anesthesia applied septoplasty operations

Exclusion Criteria:

Patients with uncontrolled hypertension, Diabetes Mellitus cerebrovascular disease, coagulopathy, morbid obesity ((BMI ≥35) and those with renal disease will not be taken

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patients that are controlled hypotensive anesthesia applied septoplasty operations
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-04-05 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Thiol / Disulfide Balance | between the start of surgery and the end of surgery (approximately 1 hour)
  Oxidative stress marker, that shows dynamic thiol-disulphide homeostasis

CONTACTS AND LOCATIONS:
Overall Officials: Leyla Kazancıoğlu, Asst. Prof., Principal Investigator — Recep Tayyip Erdoğan University Medical School Department of Anesthesia
Locations (1):
- Recep Tayyip Erdogan University Training and Research Hospital, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No